CLINICAL TRIAL: NCT00971763
Title: A Phase II Multicentre Trial of Gemcitabine, CVP, and Rituximab (R-GCVP) for the Treatment of Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma, Considered Unsuitable for R-CHOP Chemotherapy
Brief Title: Gemcitabine Hydrochloride, Cyclophosphamide, Vincristine Sulfate, Prednisolone, and Rituximab in Treating Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000644293; UCL/05/154 (Other: University College London); 2005-003888-23 (EudraCT Number); EU-20951
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2009-09

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Gemcitabine; Prednisolone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-GCVP (Experimental): Up to 6 x 21 day cycles of R-GCVP:
  * Gemcitabine 750mg/m^2 days 1 & 8 (increasing to 875mg/m^2 for cycle 2 & 1g/m^2 for subsequent cycles if tolerated satisfactorily)
  * Cyclophosphamide 750mg/m^2 day 1
  * Vincristine 1.4mg/m^2 day 1 (capped at 2mg)
  * Prednisolone 100mg/day days 1-5
  * Rituximab 375mg/m^2 day 1
  * Neulasta 6mg day 9
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: gemcitabine hydrochloride; Drug: prednisolone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: gemcitabine hydrochloride
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride, cyclophosphamide, vincristine sulfate, and prednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving more than one drug (combination chemotherapy) together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying giving gemcitabine hydrochloride, cyclophosphamide, vincristine sulfate, and prednisolone together with rituximab to see how well it works in treating patients with newly diagnosed diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether rituximab, in combination with non-cardiotoxic chemotherapy comprising gemcitabine hydrochloride, cyclophosphamide, vincristine sulfate, and prednisolone, is efficacious in a group of patients who are unfit for CHOP chemotherapy.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8; cyclophosphamide IV, vincristine sulfate IV, and rituximab IV on day 1; and oral prednisolone once daily on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20-positive diffuse large B-cell non-Hodgkin lymphoma (DLBCL) according to the current WHO classification, including all morphological variants

  * Newly diagnosed disease
  * Bulky stage IA-IV disease

    * No non-bulky stage IA disease
* Measurable disease
* Not eligible for CHOP chemotherapy due to impaired cardiac function

  * Cardiac status that does not allow the administration of 8 courses of R-CHOP chemotherapy, as defined by 1 of the following criteria:

    * Ejection fraction less than 50% as assessed by either ECHO or MUGA scan
    * NYHA class III-IV
* No high-grade transformation of low-grade lymphoma
* No symptomatic central nervous system or meningeal involvement by the lymphoma
* No AIDS-related lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 3 months
* Platelet count > 100 x 10^9/L
* WBC > 3 x 10^9/L
* Neutrophils > 1.5 x 10^9/L (unless elevated level attributed to bone marrow infiltration by lymphoma)
* Serum bilirubin < 50 μmol/L
* Transaminases < 2.5 times upper limit of normal (unless elevated level attributed to lymphoma)
* Glomerular filtration rate > 30 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent uncontrolled medical condition
* No active malignant disease, other than non-melanotic skin cancer or carcinoma in situ of the uterine cervix, within the past 10 years
* No positive serology for HIV
* No medical or psychiatric conditions that compromise the patient's ability to give informed consent

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or other investigational drug for this indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | End of treatment

SECONDARY OUTCOMES:
Toxicity | End of treatment
Progression-free survival | Not specified in protocol
Overall survival | Not specified in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fields, MD, Principal Investigator — Cancer Research UK
Locations (4):
- United Kingdom (4):
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Leeds General Infirmary, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Cancer Research UK and University College London Cancer Trials Centre, London, England

REFERENCES:
- [Derived] Fields PA, Townsend W, Webb A, Counsell N, Pocock C, Smith P, Jack A, El-Mehidi N, Johnson PW, Radford J, Linch DC, Cunnningham D. De novo treatment of diffuse large B-cell lymphoma with rituximab, cyclophosphamide, vincristine, gemcitabine, and prednisolone in patients with cardiac comorbidity: a United Kingdom National Cancer Research Institute trial. J Clin Oncol. 2014 Feb 1;32(4):282-7. doi: 10.1200/JCO.2013.49.7586. Epub 2013 Nov 12. PMID 24220559